CLINICAL TRIAL: NCT01218425
Title: Dopaminergic Modulation of Cognition and Psychomotor Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 10-3-056
Record Dates: First submitted 2010-09-22; First posted 2010-10-11 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Dopamine Activity; Episodic Memory Consolidation; Response Preparation
Keywords: dopamine; EEG; episodic memory; contingent negative variation; response preparation; levodopa; methylphenidate
MeSH Terms: interventions — Methylphenidate; Levodopa; Carbidopa; Domperidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Medication (Experimental): In this study, a crossover design is applied. All participants receive all three treatments in randomized order on separate days.
  Interventions: Drug: Methylphenidate 40 mg; Drug: Levodopa/carbidopa 125 mg; Drug: Domperidon 10 mg

INTERVENTIONS:
Drug: Methylphenidate 40 mg — Oral dose 40 mg
  Other Names: Ritalin RVG 03957
Drug: Levodopa/carbidopa 125 mg — oral dose, 100 mg levodopa, 25 mg carbidopa in one capsule
  Other Names: Sinemet RVG08740
Drug: Domperidon 10 mg — Domperidon 10 mg
  Other Names: Domperidon RVG 23565

SUMMARY:
A recent study at our lab showed increased episodic memory consolidation and response readiness after treatment with methylphenidate in healthy volunteers. The investigators seek to replicate and extend these findings. Furthermore the pharmacological specificity of these effects will be studied. Since methylphenidate has an effect on two neurotransmitters, dopamine and noradrenaline, either could be responsible for the observed effects. In order to explore the dopaminergic contribution to this effect, the study proposed here includes not only methylphenidate but also levodopa/carbidopa, which only affects dopamine and not noradrenaline.

In this study, 20 healthy males and females between 18 and 45 years of age will participate. They will be recruited via advertisements at Maastricht University and in local newspapers.

Participants will be treated once with methylphenidate, once with levodopa/carbidopa and once with placebo. All medications will be administered orally with a capsule.

It is hypothesized that methylphenidate and levodopa/carbidopa will both enhance episodic memory consolidation and improve response readiness

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 to 45 years of age
* Healthy (i.e. absence of all exclusion criteria), normal static binocular acuity (corrected or uncorrected),
* Body mass index between 18.5 and 30
* Willingness to sign an informed consent.

Exclusion Criteria:

* history of cardiac, hepatic, renal, pulmonary, neurological, gastrointestinal, haematological or psychiatric illness.
* history of depression, bipolar disorder, anxiety disorder, panic disorder, psychosis, or attention deficit hyperactivity disorder will be excluded from participation.
* first-degree relative with a psychiatric disorder or a history with a psychiatric disorder
* excessive drinking (>20 glasses of alcohol containing beverages a week
* pregnancy or lactation
* use of medication other than oral contraceptives
* use of recreational drugs from 2 weeks before until the end of the experiment
* any condition in which gastrointestinal motility might carry any risk
* any sensory or motor deficits which could reasonably be expected to affect test performance

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Behavioral score on the Word learning test | 1 day
  Number of words recalled in the word learning test

SECONDARY OUTCOMES:
CNV amplitude | 1 day
  Amplitude of the CNV wave in the EEG
Reaction time on the CNV | 1 day
  Reaction time in the response preparation task in which CNV is measured

CONTACTS AND LOCATIONS:
Overall Officials: Eric Vuurman, Dr., Principal Investigator — Dept Neuropsychology and Psychopharmacology, Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands